CLINICAL TRIAL: NCT00900302
Title: Study of The Examination of Sentinel Lymph Nodes for OX-40 Expression in Patients With Cancer
Brief Title: OX-40 Protein Expression in the Sentinel Lymph Nodes of Patients With Cancer
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000443230; P30CA069533 (NIH); OHSU-1085; OHSU-SOL-05045-L
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific; squamous cell carcinoma of the anus; squamous cell carcinoma of the bladder; squamous cell carcinoma of the esophagus; squamous cell carcinoma of the gallbladder; squamous cell carcinoma of the skin; squamous cell carcinoma of the vulva; squamous cell lung cancer; vaginal squamous cell carcinoma; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage I verrucous carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; stage I squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; squamous cell carcinoma of unknown primary; cervical squamous cell carcinoma; penile squamous cell carcinoma; recurrent anal cancer; stage I anal cancer; stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; stage IV anal cancer; recurrent bladder cancer; stage I bladder cancer; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer; recurrent esophageal cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; localized gallbladder cancer; recurrent gallbladder cancer; unresectable gallbladder cancer; recurrent vulvar cancer; stage I vulvar cancer; stage II vulvar cancer; stage III vulvar cancer; stage IV vulvar cancer; recurrent cervical cancer; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent skin cancer; newly diagnosed carcinoma of unknown primary; recurrent carcinoma of unknown primary; recurrent penile cancer; stage I penile cancer; stage II penile cancer; stage III penile cancer; stage IV penile cancer; recurrent melanoma; stage IA melanoma; stage IB melanoma; stage IIA melanoma; stage IIB melanoma; stage IIC melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma; stage IV melanoma
MeSH Terms: conditions — Neoplasms; Breast Neoplasms, Male; Breast Neoplasms; Anus Neoplasms; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms; Urinary Bladder Neoplasms; Esophageal Neoplasms; Gallbladder Neoplasms; Vulvar Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Skin Neoplasms; Neoplasms, Unknown Primary; Penile Neoplasms; Melanoma | interventions — Immunohistochemistry; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: protein expression analysis — The first ten cases will be reviewed to assess the spectrum of OX-40 expression and to devise a semiquantitative scoring system. Each slide will be scanned in its entirety and then scored according to representative views with the greatest expression of immunostaining. Two independent viewers, who will be blinded to clinical data and outcome at the time of scoring, will review all slides. Scores from these independent readings will be compared, and differences were resolved upon mutual review of given cases. We will estimate the distribution of OX-40 IHC score by tumor type and tumor stage. OX-40 IHC score will be correlated with the IHC scores of other markers using Spearman's correlation coefficient. Kruskal-Wallis test will be used to test whether OX-40 IHC score is comparable between tumor type and tumor stage
Other: immunohistochemistry staining method — 5-micron sections will be cut, mounted on capillary gap slides and dried in a 60°C oven. The slides will then be then deparaffinized in xylene baths and gradually hydrated in graded alcohol. For epitope retrieval, the slides are placed in baths of 0.5 M Tris buffer at pH 10 and subjected to microwave irradiation for at least 19 minutes. The slides will be cooled and washed with deionized water and 0.05% TWEEN. They are then placed in a blocking solution of 0.3% bovine serum albumin, drained, and placed in wells of their primary antibody in a humidity chamber at room temperature overnight. Primary mouse antihuman antibodies will include anti-OX-40, anti-CD4, and anti-HLA class II. Anti-rat CD45 will be used as a negative control for each section. The slides will then be then washed and placed in their appropriate biotinylated anti-mouse secondary antibody for 24 minutes. Endogenous peroxidase in the samples is blocked using a solution of 3% hydrogen peroxide.
Other: laboratory biomarker analysis — Lymphocytes will be collected from fresh tissue and peripheral blood (PBLs) for use in marker analysis and in vitro assays of immune function. Tissues will be dissociated to obtain lymphocytes
Procedure: biopsy — De-identified tissue samples will be obtained from the OHSU Pathology Department. Tissues will consist of paraffin blocks collected either prospectively for previous cases, or fresh tissue collected prospectively for patients enrolled in the study. For either case, tissue will be collected only after tissue necessary for the adequate rendering of the pathologic diagnosis has been collected by the pathology Department. Thus, the collection of tissue will not compromise patient diagnosis/care.

SUMMARY:
RATIONALE: Studying protein expression in sentinel lymph node tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help the study of cancer in the future.

PURPOSE: This laboratory study is evaluating OX-40 protein expression in the sentinel lymph nodes of patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the qualitative and quantitative expression of OX-40 and related markers in sentinel lymph nodes previously removed from patients with cancer.
* Determine the qualitative and quantitative expression of OX-40 and related markers in sentinel lymph nodes freshly removed from patients with cancer.
* Correlate the expression of OX-40 and related markers in sentinel lymph node tissue with expression in nonsentinel tissue from primary tumors and nonsentinel lymph nodes, tumor stage, and patient outcomes.

OUTLINE: Sections of primary tumors, nonsentinel lymph nodes, and sentinel lymph nodes will be analyzed for expression of OX-40 by immunohistochemistry. Sections of negative (no tumor metastases) lymph nodes will be used as internal controls. Fresh tissue and blood will be tested for marker analysis and in vitro assays of immune function.

PROJECTED ACCRUAL: A total of 100 specimens from sentinel lymph nodes previously removed from cancer patients and 100 specimens from sentinel lymph nodes freshly removed from cancer patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed cancer, including, but not limited to, the following:

  * Melanoma
  * Breast cancer
  * Invasive squamous cell cancer
  * Other cancers for which patients underwent or will undergo the following:

    * Adequate archived paraffin-embedded tissue for making slides for immunostaining
    * Adequate freshly removed sentinel lymph node (and primary tumor, if available) tissue for laboratory assays
* Clinical data and date of last follow-up on tumor stage and status must be available
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: De-identified tissue samples will be obtained from the OHSU Pathology Department
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2005-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
OX-40 expression | During immunostaining
  The first ten cases will be reviewed to assess the spectrum of OX-40 expression and to devise a semiquantitative scoring system. Each slide will be scanned in its entirety and then scored according to representative views with the greatest expression of immunostaining
Disease-free survival | During data analysis
  Kaplan-Maier method will be used to estimate the disease-free survival, and a log-rank test will be used to compare the disease-free survival between high vs. low OX-40 groups

CONTACTS AND LOCATIONS:
Overall Officials: John T. Vetto, MD, FACS, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States